CLINICAL TRIAL: NCT06764953
Title: A Randomized Controlled Clinical Trial Evaluating The Efficacy of an Amnion Membrane Allograft Intended for Use in the Management of Non- Healing Venous Leg Ulcers Versus Standard Of Care Alone
Brief Title: Clinical Trial Evaluating an Amnion Membrane Allograft Intended for Use in the Management of Non- Healing Venous Leg Ulcers Versus Standard Of Care Alone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skye Biologics Holdings, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKY-WP-VLU-02
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Venous Leg Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SOC primary dressing with E-GRAFT ™ (Experimental): Participants receive standard of care with E-GRAFT™
  Interventions: Other: E-GRAFT ™
- SOC primary dressing with FIBRACOL™ (Active Comparator): Participants receive standard of care with FIBRACOL™
  Interventions: Device: FIBRACOL™

INTERVENTIONS:
Other: E-GRAFT ™ — E-GRAFT™ that is a dehydrated thick amniotic allograft processed and approved for use as a Human Cellular and Tissue-Based Product (HCT/P) under FDA 21 CFR 1271 and Section 361 of the Public Health Service (PHS) Act.
  Arms: SOC primary dressing with E-GRAFT ™
Device: FIBRACOL™ — 510K FDA cleared Collagen alginate dressing
  Arms: SOC primary dressing with FIBRACOL™

SUMMARY:
The main purpose of this research study is to compare the proportion of wound closure in subjects that receive E-GRAFT™ with SOC versus FIBRACOL™ with SOC. Other research purposes include the following:

* Rate of wound closure
* Change in ulcer size over 12 weeks
* Any adverse events or reactions (side effects)
* Change in pain levels
* Occurrence of infection

DETAILED DESCRIPTION:
The purpose of this clinical evaluation is to collect patient outcome data on a commercially available E-GRAFT™ that is a dehydrated thick amniotic allograft processed and approved for use as a Human Cellular and Tissue- Based Product (HCT/P) under FDA 21 CFR 1271 and Section 361 of the Public Health Service (PHS) Act. In this trial, two groups of Venous Leg Ulcers (VLUs) will receive standard of care (SOC) treatment for their condition. Half of the patients will receive a 510K FDA cleared Collagen alginate dressing FIBRACOL™ and the other half will have E-GRAFT™ dehydrated tissue allograft as the primary dressing. The primary endpoint is the percentage of patients that go on to complete closure of the target ulcer between the two groups: SOC with FIBRACOL™ or SOC with E-GRAFT™. Secondary endpoints include the proportion of subjects achieving complete wound closure of the target ulcer by the end of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older.
2. At randomization subjects must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 20.0 cm2 measured post debridement with manual measure.
3. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
4. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
5. The subject must consent to using the prescribed off-loading method for the duration of the study.
6. The subject must agree to attend the weekly study visits required by the protocol.
7. The subject must be willing and able to participate in the informed consent process.
8. The target ulcer must be full thickness on the foot or leg that does not probe to bone.
9. Adequate circulation to the affected foot as documented by any of the following methods performed within 3 months of the first screening visit:

   1. TCOM ≥30 mmHg
   2. ABI between 0.7 and 1.3
   3. PVR: Biphasic
   4. TBI ˃0.6
   5. As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle
10. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
11. Target ulcers must have been treated with compression therapy for at least 14 days prior to randomization.

Exclusion Criteria:

1. A subject known to have a life expectancy of < 6 months is excluded.
2. If the target ulcer is infected or if there is cellulitis in the surrounding skin, the subject is excluded.
3. Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
4. Index ulcer and/or index ulcer limb may have had prior infection(s), but infection(s) must be adequately treated and controlled
5. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
6. The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
7. A subject with a previous partial amputation on the affected leg is excluded if the resulting deformity impedes proper offloading of the target ulcer.
8. If a subject is diabetic and has a glycated hemoglobin (HbA1c) greater than or equal to 12% taken at or within 3 months of the initial screening visit he/she is excluded.
9. If a subject has a serum creatinine ≥ 3.0mg/dL within 6 months of randomization he/she is excluded.
10. The subject is excluded if the surface area measurement of the target ulcer has reduced in size by more than 30% in the 2 weeks prior to the initial screening during the 2-week screening phase: the 2 weeks from the initial screening visit (SV1) to the TV1/randomization visit during which time the subject received SOC.
11. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
12. A potential subject with end stage renal disease requiring dialysis is excluded.
13. A subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
14. A subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit is excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of index ulcers "healed" at 12 weeks | 12 weeks
  Investigator assessment of healing (100% epithelization w/no drainage), measurements of ulcer size using manual measurements

SECONDARY OUTCOMES:
Time to healing within 12 weeks | 12 weeks
  Time to healing will be taken as the time of first assessment (i.e. before confirmation within two weeks) of complete healing.
Percentage Area Reduction over 12 week period | 12 weeks
  Digital imaging

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Zelen, DPM FACFAS, Principal Investigator — Professional Education and Research Institute
Locations (1):
- Professional Education and Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No